CLINICAL TRIAL: NCT03803852
Title: Rotation of Hydrophobic Acrylic Lenses - Rayner RA0800C & Alcon Clareon & Hoya Nanex & Hoya Vivinex XY1-EM & RayOne EMV Toric & PODEYE Toric
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Ao.Univ.Prof.Dr. Rupert Menapace, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1978/2018
Record Dates: First submitted 2019-01-07; First posted 2019-01-15 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Age Related Cataracts; Astigmatism
MeSH Terms: conditions — Astigmatism | interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Intervention Model Description: The study involves 5 different groups. All groups will be investigated seperately.
  Alcon Clareon toric group: 130 eyes Rayner RayOne group: 130 eyes Hoya Nanex group: 130 eyes Hoya Vivinex Impress: 120 eyes Rayner RayOne EMV toric group: 120 eyes PODEYE Toric: 120 eyes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 0° (Experimental): Implantation of an intraocular lens Rayner RayOne or Hoya Nanex or Hoya Vivinex Impress on axis 0°
  Interventions: Device: Intraocular Lens Implantation
- 45° (Experimental): Implantation of an intraocular lens Rayner RayOne or Hoya Nanex or Hoya Vivinex Impresson axis 45°
  Interventions: Device: Intraocular Lens Implantation
- 90° (Experimental): Implantation of an intraocular lens Rayner RayOne or Hoya Nanex or Hoya Vivinex Impress on axis 90°
  Interventions: Device: Intraocular Lens Implantation
- 135° (Experimental): Implantation of an intraocular lens Rayner RayOne or Hoya Nanex or Hoya Vivinex Impresson axis 135°
  Interventions: Device: Intraocular Lens Implantation

INTERVENTIONS:
Device: Intraocular Lens Implantation — Implantation of an intraocular lens Rayner RayOne or Hoya Nanex or Hoya Vivinex Impressinto the capsular bag using an injector, after removing of the human cristalline lens.
  Implantation of the Alcon Clareon toric and Rayner RayOne EMV toric IOL and PODEYE Toric IOL on the axis according to the steep meridian of the cornea

SUMMARY:
The investigational devices are approved intraocular lenses (IOL) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. Within the study, three different IOLs will be investigated and separately evaluated. Cataract surgery with IOL implantation will be performed in subjects who have signed an informed consent form. Postoperative examinations will be postoperative refraction, visual acuity, slitlamp examination, and rotation of the IOL within 1 hour, 1 week, 1 month and 4-7 months.

In the Alcon Clareon toric, RayOne EMV toric and PODEYE Toric group, patients receive a toric IOL according to their preoperative astigmatism

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral age-related cataract necessitating phacoemulsification extraction and posterior IOL implantation
* Age: 45 to 95
* Need for spherical IOL correction between 10.00 and 30.00 D
* Need for spherical IOL correction between +6.00 and +30.00 D (Alcon Clareon toric group)
* Need for spherical IOL correction between +10.00 and +25.00 D (Rayner RayOne EMV toric group)
* Preoperative pupil dilation in mydriasis ≥ 7.0 mm (Hoya, Rayner groups)
* Astigmatism of at least 1.0 Diopters (Alcon Clareon toric and Rayner RayOne EMV toric groups and PODEYE Toric)
* Pupil dilation >5.5mm (Alcon Clareon toric Rayner RayOne EMV toric group)

Exclusion Criteria:

* Preceding ocular surgery or trauma

  * Recurrent intraocular inflammation of unknown etiology
  * Uncontrolled glaucoma
  * Uncontrolled systemic or ocular disease
  * Blind fellow eye
  * Microphthalmus
  * Corneal abnormality (Corneal scaring)
  * History of uveitis/iritis
  * Iris neovascularization
  * Proliferative diabetic retinopathy
  * Pregnancy
  * Lactation
  * Females of childbearing age will be asked if pregnancy is possible

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change of axial intraocular lens position | 7 months
  Change in axis position of an intraocular lens Rayner RayOne or Hoya Nanex or Hoya Vivinex Impress or Alcon Clareon toric or Rayner RayOne EMV toric or PODEYE Toric from end of surgery (baseline axis) to 1 hour, 1 week, 1 month and 4-7 months (end of study visit). The change in axis position will be evaluated with respect to the baseline measurement at the end of surgery. Differences in axis position will be described as rotation in degrees (0 to 360°)

SECONDARY OUTCOMES:
Decentration | 7 months
  Decentration of the intraocular lens Rayner RayOne or Hoya Nanex or Hoya Vivinex Impress or Alcon Clareon toric or Rayner RayOne EMV toric or PODEYE Toric will be measured with the Casia 2 OCT. Decentration will be described as "Decentration in milimeter"
Tilt | 7 months
  Tilt of the intraocular lens Rayner RayOne or Hoya Nanex or Hoya Vivinex Impress or Alcon Clareon toric or Rayner RayOne EMV toric or PODEYE Toric will be measured with the Casia 2 OCT. Tilt will be described as "Tilt in degrees at a certain axis"
Anterior chamber depth | 1 month
  The anterior chamber depth (Axial position of the IOL) of the intraocular lens Rayner RayOne or Hoya Nanex or Hoya Vivinex Impress or Alcon Clareon or Rayner RayOne EMV toric or PODEYE Toric will be measured with the Casia 2 OCT after 1 month. The anterior chamber depth will be measured in milimeter
Best corrected visual acuity (BCVA) | 7 months
  BCVA will be measured at 1 week, 1 month and 4 to 7 months. The BCVA will be described as the minimum angle of resolution (logMar)
UCIVA in the Alcon Clareon toric and Rayner RayOne EMV toric groups | 7 months
  Uncorrected Intermediate Visual Acuity mono or bilateral

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Menapace, Prof.Dr., Principal Investigator — Medical University Vienna
Locations (1):
- Medical University of Vienna Allgemeines Krankenhaus, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schartmuller D, Lisy M, Mahnert N, Schranz M, Danzinger V, Schwarzenbacher L, Pieh S, Abela-Formanek C, Leydolt C, Menapace R. Rotational stability and refractive outcomes of a new hydrophobic acrylic toric intraocular lens. Eye Vis (Lond). 2024 Jul 2;11(1):25. doi: 10.1186/s40662-024-00393-2. PMID 38951940